CLINICAL TRIAL: NCT06520254
Title: The Effectiveness of Massage in Pain Reduction and Its Influence on the Range of Motion (ROM) of the Shoulder Complex in Patients With Shoulder Pain in Primary Care
Brief Title: The Effectiveness of Massage Therapy in Patients With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Kassolik, Phd, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pain in shoulder
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, parallel, two-arm trial
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): Participants in the massage group will receive 6 massage sessions (twice a week for 3 weeks).
  Interventions: Other: Massage therapy
- Control group (No Intervention): Participants in the control group will receive 2 massage sessions, first one at the baseline, second one after 3 weeks.

INTERVENTIONS:
Other: Massage therapy — A 30-minute massage session will be applied in the following structures:
  * Flexor hallucis longus muscle,
  * Flexor digitorum longus muscle,
  * Tibialis posterior muscle,
  * Semitendinosus muscle,
  * Semimembranosus muscle,
  * Gluteus maximus muscle,
  * Longissimus muscle,
  * Levator costarum muscles 1-5 During the massage session basic Swedish massage techniques were used.
  Arms: Massage group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of massage in pain reduction and its influence on the range of motion of the shoulder complex in SP.

The main questions it aims to answer are:

1. Does normalizing tissue tension through massage therapy in the intercostal nerve entrapment mechanism reduce pain in the shoulder area?
2. Does normalizing tissue tension through massage therapy in the intercostal nerve entrapment mechanism increase the range of motion of the shoulder complex?

Researchers will compare a dedicated massage protocol to a control group to see if the massage protocol works to treat shoulder pain.

Participants in the massage group will:

Take part in 6 massage sessions (twice a week for 3 weeks) in the

Participants in the control group will:

Take part in 2 massage sessions (after the first and second assessment)

DETAILED DESCRIPTION:
The aim of the study was to evaluate the effectiveness of massage therapy based on tensegrity principle in pain reduction and its influence on the range of motion of the shoulder complex in shoulder pain. .

Eesearch questions:

1. Does the normalization of the tension of the tissues involved in the intercostal nerve entrapment mechanism reduce pain in the shoulder area?
2. Does the normalization of the tension of the tissues involved in the intercostal nerve entrapment mechanism increase the range of motion of the shoulder complex?
3. Does the intercostal nerve entrapment affect the pressure sensitivity of the muscles including the shoulder complex?89
4. What potential mechanisms may be induced by tensegrity massage in diseases of the shoulder complex?

Patients with symptoms of shoulder pain will be recruited for the study by general practitioners.

The following parameters related to the function of shoulder will be assessed:

1. The active range of flexion, abduction and extension-adduction-rotation (hand behind back) of the upper limb were assessed.
2. Pain sensations by the visual analogue scale-VAS
3. The functional status of the shoulder complex by the UCLA scale (The University of California at Los Angeles Shoulder Score).
4. Pain treshold by an algometer, the pressure

The study will rely on the palpation assessment and the massage methodology described in the recommendations of the Polish Society of Physiotherapy, Polish Society of Family Medicine and College of Family Physicians in Poland.

ELIGIBILITY:
Inclusion Criteria:

* age over 40 years,
* written consent to participate in the study,
* pain in the shoulder girdle area lasting at least 3 months,
* no medical contraindication of massage therapy;

Exclusion Criteria:

* Injuries, congenital defects in the chest area, cancer, deep vein thrombosis, heart attack in the last 5 years,
* Presence of inflammatory conditions in the respiratory, digestive, and genitourinary systems

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in the pain threshold of the shoulder after therapy compared to baseline | 1) baseline, 2) 3 weeks after the first massage session massage session
  Measuring device: The Wagner FPXTM Algometer produced by The Wagner Instruments, Greenwich CT, USA, Change = (Value after therapy - baseline)
Change in the The University of California at Los Angeles Shoulder Score after therapy compared to baseline | 1) baseline, 2) 3 weeks after the first massage session massage session
  Measuring device: UCLA scale (The University of California at Los Angeles Shoulder Score) , Change = (Value after therapy - baseline)

SECONDARY OUTCOMES:
Change in the Visual analog scale score after therapy compared to baseline | 1) baseline, 2) 3 weeks after the first massage session massage session
  Measuring device: VAS scale - Visual analog scale - a continuous scale comprised of a horizontal line, 100 mm in length, anchored by "no pain" (score of 0) and "worst imaginable pain" score of 10, Change = (Value after therapy - baseline)
Change in ROM after therapy compared to baseline | 1) baseline, 2) 3 weeks after the first massage session massage session
  Measuring device: a goniometr, Change = (Value after therapy - baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Dobrzycka, Phd, Principal Investigator — Idependent researcher
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Artus M, Holt TA, Rees J. The painful shoulder: an update on assessment, treatment, and referral. Br J Gen Pract. 2014 Sep;64(626):e593-5. doi: 10.3399/bjgp14X681577. No abstract available. PMID 25179075
- [Result] Kassolik K, Jaskolska A, Kisiel-Sajewicz K, Marusiak J, Kawczynski A, Jaskolski A. Tensegrity principle in massage demonstrated by electro- and mechanomyography. J Bodyw Mov Ther. 2009 Apr;13(2):164-70. doi: 10.1016/j.jbmt.2007.11.002. Epub 2007 Dec 21. PMID 19329052